CLINICAL TRIAL: NCT06970483
Title: Comparison of the Efficacy of Sublingual Misoprostol and Intravenous Tranexamic Acid for Postpartum Hemorrhage Prophylaxis in Cesarean Delivery
Brief Title: Comparison of the Efficacy of Misoprostol and Tranexamic Acid for Postpartum Hemorrhage Prophylaxis in Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Ağbal, Clinical Doctor, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK1-2023-774
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Postpartum Hemorrhage; Cesarean Section Complications; Delivery Complication
Keywords: postpartum hemmorrhage; ceserean section; maternal complications of delivery; prostoglandine1; tranexamic asid
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Tranylcypromine; Misoprostol; Tablets

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group 1 received tranexamic acid (Transamin 10% ampoule, 2.5 mL / 250 mg, Actavis Pharmaceuticals, Turkey); 1 gram was administered intravenously during the lower segment incision.
  In addition,patients received 20 International Units (IU) of oxytocin (Synpitan Forte, 5 IU/mL ampoule I.M./I.V., Deva Holding A.Ş., Turkey).
  Interventions: Drug: Tranexamic acid
- Group 2: Group 2 received misoprostol (Cytotec, 200 mcg tablet, Pfizer Inc., USA); 400 mcg were administered sublingually immediately after delivery of the baby and clamping of the umbilical cord.
  In addition,patients received 20 IU of oxytocin (Synpitan Forte, 5 IU/mL ampoule I.M./I.V., Deva Holding Inc., Turkey).
  Interventions: Drug: Misoprostol 200mcg Tab
- Group 3 control group: Group 3 received only 20 IU of oxytocin (Synpitan Forte, 5 IU/mL ampoule I.M./I.V., Deva Holding Inc., Turkey). No additional pharmacological agents were administered to this group.

INTERVENTIONS:
Drug: Tranexamic acid — Transamine1 gram was administered intravenously during the lower segment incision.
  Other Names: Transamine 10% ampoule, 2.5 mL / 250 mg
  Groups: Group 1
Drug: Misoprostol 200mcg Tab — Cytotec 400 micrograms were administered sublingually immediately after delivery of the baby and clamping of the umbilical cord.
  Other Names: Cytotec 200 Mcg Tablet
  Groups: Group 2

SUMMARY:
Postpartum hemorrhage (PPH) is an obstetric emergency, with an estimated incidence ranging from 2.8% to 7.9%. Recent studies indicate an increasing trend in the frequency of PPH.Although it is more commonly seen in developing countries, it remains a significant cause of maternal morbidity and mortality worldwide. Therefore, early diagnosis and prompt, accurate intervention are critically important.

Despite the rising incidence of PPH, maternal mortality rates have declined. This improvement is largely attributed to better identification of risk factors, timely diagnosis, and effective intervention.

To prevent PPH globally, active management of the third stage of labor has been widely implemented. This approach includes the use of pharmacologic agents, uterine massage, and controlled traction for placental delivery.Among pharmacological agents, the most commonly used include oxytocin, ergot alkaloids (e.g., ergometrine), tranexamic acid, prostaglandin E1 (misoprostol), prostaglandin F2α, and oxytocin analogues (e.g., carbetocin).Oxytocin is the most widely used agent for PPH prophylaxis.

The aim of this study is to compare the efficacy of tranexamic acid and misoprostol in the prophylaxis of postpartum hemorrhage.

DETAILED DESCRIPTION:
The study included emergency or elective cases scheduled for cesarean delivery at the Obstetrics and Gynecology Clinic, Maternity Ward of Etlik City Hospital, between December 2023 and December 2024.

Patients were divided into three groups. Group 1 received tranexamic acid (Transamin 10% ampoule, 2.5 mL / 250 mg, Actavis Pharmaceuticals, Turkey); 1 gram was administered intravenously (I.V.) during the lower segment incision.

Group 2 received misoprostol (Cytotec, 200 mcg tablet, Pfizer Incorporated company (Inc. , USA); 400 micrograms(mcg) were administered sublingually immediately after delivery of the baby and clamping of the umbilical cord.

In addition, all patients received 20 International Units (IU) of oxytocin intramuscularly (I.M.) (Synpitan Forte, 5 IU/mL ampoule I.M./I.V., Deva Holding Inc. , Turkey).

Despite the medical treatments administered, in cases where hemorrhage developed intraoperatively or postoperatively, additional interventions were performed, including medical (additional doses of oxytocin/tranexamic acid/misoprostol), mechanical (Bakri balloon), or surgical methods (uterine artery/hypogastric artery ligation, B-Lynch/Hayman sutures, postpartum hysterectomy).

The parameters to be examined in the research are as follows:

1. Patients' postoperative 1st, 2nd, and 6th-hour vital signs (pulse rate, systolic and diastolic blood pressure, temperature, oxygen saturation).
2. Shock indices.
3. Hemogram and hematocrit values at 6-24 hours postoperatively.
4. Duration of the surgery.
5. Adverse effects experienced by the patients.
6. Additional treatments administered.
7. Whether blood transfusion was performed or not. In this study, the G-power analysis program was used to determine the minimum sample size, taking into account a 10% margin of error. According to the analysis results, the minimum number of patients to be included in the study for a total of 75 patients across 3 groups was determined. Statistical analysis of the data obtained in the study will be conducted using the Statistical Package for the Social Sciences (SPSS) version 22 software package. A 95% confidence interval will be calculated for each variable, and results will be considered statistically significant for p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-45 years
* gestational age between 37 and 41 weeks
* Perfomed ceserean section for delivery

Exclusion Criteria:

* did not provide informed consent,
* with comorbidities (such as heart, liver, or lung diseases),
* high-risk pregnancy (e.g., intrauterine growth restriction, cholestasis, preeclampsia, eclampsia, multiple pregnancies)
* known allergies to tranexamic acid or misoprostol
* known coagulation disorders

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — women
Study Population: The study included emergency or elective cases scheduled for cesarean delivery at the Obstetrics and Gynecology Clinic, Maternity Ward of Etlik City Hospital, between December 2023 and December 2024
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Comparison of patients' preoperative and postoperative hemogram levels | 24 hours
  Hemogram values were compared at 0-24 hours postoperatively
Comparison of patients' preoperative and postoperative hematocrit levels | 24 hours
  Hematocrit values were compared at 0-24 hours postoperatively
Comparison of patients' postoperative shock indices | 24 hours
  postoperative shock indices were compared at 0-24 hours postoperatively

SECONDARY OUTCOMES:
Comparison of the patients' postoperative heart rate | 24 hours
  postoperative heart rates were compared at 0-24 hours postoperatively
Comparison of the patients' postoperative systolic and diastolic blood pressure | 24 hours
  postoperative systolic and diastolic blood pressures were compared at 0-24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Turkey (Türkiye)